CLINICAL TRIAL: NCT04657471
Title: Hospitalization or Outpatient ManagEment of Patients With Suspected or Confirmed SRAS-CoV-2 Infection: the Revised HOME-CoV Score Study.
Brief Title: Hospitalization or Outpatient ManagEment of Patients With SRAS-CoV-2 Infection - Revised HOME-CoV Score Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-A03067-32
Record Dates: First submitted 2020-12-06; First posted 2020-12-08 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2020-12

CONDITIONS: Coronavirus Infection
Keywords: Outpatients; COVID-19; Risk assessment model; home treatment
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Intervention Model Description: Multicentre prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- revised HOMe-CoV (Experimental): Revised HOME-CoV
  Interventions: Other: revised HOME-CoV score

INTERVENTIONS:
Other: revised HOME-CoV score — Educational lectures, posters, and pocket cards showing and explaining the revised HOME-CoV score are communicated to participating Emergency Departments.
  For included patients, the physician-in-charge calculates the revised HOME-CoV. Patients with a score <2 qualified for home treatment. They qualified otherwise for hospitalization. For patients with a score > 4, hospitalization in a unit allowing monitoring of vital parameters is recommended. However, the physician-in-charge can overrule the qualification for home treatment or for hospitalization in case of major medical or social reasons. A justification explaining the cause of overruling is required.

SUMMARY:
In the context of COVID-19 pandemic, identifying low-risk patients who can be safely treated at home and high-risk patients requiring hospitalization or even intensive care is crucial for Emergency Departments. Thanks to a consensus of experts using the Delphi method, we previously defined the HOME-CoV rule. The HOME-CoV rule consists of 8 items precluding home treatment for patients consulting in the Emergency Department (ED) with confirmed or highly suspected mild to moderate COVID-19. It has been validated in a prospective study, patients with a negative rule having a very-low rate of invasive ventilation or death within the 7 days following ED presentation (HOME-CoV study, NCT: 02811237).

Using logistic regression, we revised the HOME-CoV rule in order to define a score allowing. The revised HOME-CoV score comprises 7 criteria and, retrospectively assessed in the database of the HOME-CoV study, it exhibits promising performances. A revised HOME-CoV score < 2 had a sensitivity of 0.93 (0.84 to 0.98), a specificity of 0.60 (0.58 to 0.61) and negative predictive value of 1.00 (0.99 to 1.00); and a score > 4 had a sensitivity of 0.41 (0.28 to 0.54), a specificity of 0.93 (0.92 to 0.94) and a positive predictive value of 0.11 (0.07 to 0.16).

The present study aims to prospectively validate the revised HOME-CoV score, firstly, in identifying a subgroup of COVID-19 patients with a low risk of evolution to severe COVID-19 and who could be safely treated at home.

For this purpose, we will perform an interventional multicentric prospective pragmatic cohort study with implementation of the revised HOME-CoV score to triage COVID-19 patients.

DETAILED DESCRIPTION:
In all participating Emergency Departments, patients with highly suspected or confirmed COVID-19 are evaluated for potential inclusion. Clinical, biological, and imaging data that may be involved in decision-making about hospitalization, including all criteria of the revised HOME-CoV score, are collected. The revised HOME-CoV score is calculated. Patients with a score <2 qualify for home treatment. They qualify otherwise for hospitalization. For patients with a score > 4, hospitalization in a unit allowing monitoring of vital parameters is recommended. The qualification for home treatment or for hospitalization can be overruled by the physician-in-charge in case of major medical or social reasons. A justification explaining the cause of overruling is required.

A phone-call follow-up is performed on Day 7 and the patients' clinical status according to the Ordinal Scale for Clinical Improvement of COVID-19 from the World Health Organization (WHO-OSCI) is collected.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years old)
* Admitted for COVID-19 infection confirmed by a positive SARS-CoV2 RT-PCR or considered probable by the physician in charge of the patient.
* Not requiring care in intensive care unit or resuscitation unit or
* No subject of a limitation decision of active therapies,
* Free informed express consent to participate in the study orally given or signed by the patient according to local legislation,
* Insurance cover according to local legislation;

Exclusion Criteria:

* Patient admitted to the emergency room for 18 hours or more,
* Patient whose follow-up on D7 is impossible, whatever the reason,
* Patient already included in the study,
* Person deprived of their liberty by judicial or administrative decision,
* Person under psychiatric care under duress,
* Person subject to a legal protection measure,
* Person unable to express consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
The safety of the revised HOME-CoV score strategy for home treatment | 7 days
  The rate of patients with evolution to severe COVID-19 within 7 days after inclusion among patients with a revised HOME-CoV score <2.
  Severe COVID-19 is defined as a WHO-OSCI≥5, i.e., high flow nasal oxygen therapy or non-invasive ventilation (5), intubation and invasive ventilation (6), other vital support (7), or all-cause death (8).
  The revised HOME-CoV score strategy will be considered as safe if the rate of patients who experienced a WHO-OSCI≥5, will be ≤0.5% with an upper limit of the 95% confidence interval ≤1%.

SECONDARY OUTCOMES:
The efficacy of the revised HOME-CoV score strategy for home treatment | 24 hours
  The rate of patients treated at home,i.e., discharged home within 24 hours following inclusion.
The applicability of the revised HOME-CoV score strategy for home treatment | 24 hours
  the rate of patients treated at home, i.e., discharged home within 24 hours following inclusion, among patients with a revised HOME-CoV score <2
The reliability of the revised HOME-CoV score strategy for home treatment | 7 days
  The rate of patients with a revised HOME-CoV score < 2 and treated at home who were not subsequently hospitalized within the 7 days following inclusion.
The predictive performances of the revised HOME-CoV score of evolution towards a COVID-19 with a WHO-OSCI≥5. | 7 days
  The rate of patients with a WHO-OSCI≥5 within the 7 days following inclusion, i.e., high flow nasal oxygen therapy or non-invasive ventilation (5), intubation and invasive ventilation (6), other vital support (7) or all-cause death (8). The following parameters will be calculated: the area under the receiving operating curve (AUROC), sensitivity, specificity, negative likelihood ratio, positive likelihood ratio, negative predictive value and positive predictive value with <2 and >4 as cutoffs.
  7 days
The predictive performances of the revised HOME-CoV score of evolution towards a COVID-19 with a WHO-OSCI≥6 | 7 days
  The rate of patients with a WHO-OSCI≥6 within the 7 days following inclusion, i.e., intubation and invasive ventilation (6), other vital support (7) or all-cause death (8).
  The following parameters will be calculated: the area under the receiving operating curve (AUROC), sensitivity, specificity, negative likelihood ratio, positive likelihood ratio, negative predictive value and positive predictive value with <2 and >4 as cutoffs.
The predictive performances of the revised HOME-CoV score of evolution towards a fatal COVID-19 | 7 days
  The rate of patients who dead within the 7 days following inclusion
  The following parameters will be calculated: the area under the receiving operating curve (AUROC), sensitivity, specificity, negative likelihood ratio, positive likelihood ratio, negative predictive value and positive predictive value with <2 and >4 as cutoffs.
Subgroup analysis in patients with confirmed COVID-19 (positive SARS-CoV2 RT-PCR) of the predictive performances of the revised HOME-CoV score | 7 days
  The rate of patients with a WHO-OSCI≥5 within the 7 days following inclusion, i.e., high flow nasal oxygen therapy or non-invasive ventilation (5), intubation and invasive ventilation (6), other vital support (7) or all-cause death (8).
  The following parameters will be calculated: the area under the receiving operating curve (AUROC), sensitivity, specificity, negative likelihood ratio, positive likelihood ratio, negative predictive value and positive predictive value with <2 and >4 as cutoffs.
The predictive performances of the revised HOME-CoV score as compared to those of other prognostic scores for COVID-19 | 7 days
  The rate of patients with a WHO-OSCI≥5 within the 7 days following inclusion, i.e., high flow nasal oxygen therapy or non-invasive ventilation (5), intubation and invasive ventilation (6), other vital support (7) or all-cause death (8).
  The following parameters will be calculated: the area under the receiving operating curve (AUROC)
Venous thrombo-embolism in COVID-19 patients (ancillary study) | 7 days
  The rate of symptomatic and objectively confirmed deep venous thromboembolism or pulmonary embolism, and of unexplained sudden death occurring within the 7 days following ED admission.

CONTACTS AND LOCATIONS:
Overall Officials: Medhi TAALBA, Principal Investigator — CHU Rouen; David DALL'ACQUA, Principal Investigator — Jacques Lacarin Hospital Center; Anyhony CHAUVIN, Principal Investigator — AP-HP Hopital Lariboisière; Emmanuel MONTASSIER, Principal Investigator — Nantes University Hospital; Christian BRICE, Principal Investigator — CH St Brieuc; Frédéric BALEN, Principal Investigator — University Hospital, Toulouse; Kasarra BEN HAMMOUDA, Principal Investigator — CH Colmar; Marc NOIZET, Principal Investigator — CHRU Mulhouse; Romain BLONDET, Principal Investigator — Ch Mont de Marsan; Mustapha SEBBANE, Principal Investigator — University Hospital, Montpellier; Pierre-Clément THIEBAUD, Principal Investigator — AP-HP Hôpital St Antoine; Marc ANDRONIKOF, Principal Investigator — AP-HP Hôpital Béclère; Esma OUMMAMAR, Principal Investigator — CH Le Mans; Laure ABENSUR VUILLAUME, Principal Investigator — CHRU Metz-Thionville; Henrinjatovo ANDRIANJAFY, Principal Investigator — Groupe Hospitalier Nord Essonne - Longjumeau; Yann-Erick CLAESSENS, Principal Investigator — CH Princesse Grace de Monaco; Pascal BISSOLOKELE, Principal Investigator — CH Libourne; Francis COUTURAUD, Principal Investigator — CHU Brest; Séverine GOSSELIN, Principal Investigator — CHU Dijon; Mathieu VIOLEAU, Principal Investigator — CH Niort; SCHMIDT Jeannot, Principal Investigator — University Hospital, Clermont-Ferrand; Henri Hani KARAM, Principal Investigator — CHU Limoges; Meïssa KARE, Principal Investigator — CH Agen; Coralie CAYEUX, Principal Investigator — CH Remiremont; Florent FREMY, Principal Investigator — AP-HP HEGP; Nicolas PESCHANSKI, Principal Investigator — CHU Rennes; Caroline SOULIE, Principal Investigator — CH Cholet; Ombeline SUSONG, Principal Investigator — GHT La Rochelle; Stéphane GENNAI, Principal Investigator — CHU REIMS; Julie PERNET, Principal Investigator — AP-HP La Pitié-Salpêtrière; Andrea PENALOZA, Principal Investigator — Cliniques Universitaires St Luc (Bruxelles); Alexandre GHUYSEN, Principal Investigator — Centre Hospitalier Universitaire de Liege; Sonja CURAC, Principal Investigator — Hôpital Erasme (Bruxelles)
Locations (1):
- CHU Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No